CLINICAL TRIAL: NCT06647641
Title: The CurePSP Genetics Program
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: CurePSP Foundation (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Director, CurePSP Center of Care, Massachusetts General Hospital
Other Study IDs: 2024P001971
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: PSP; PSP - Progressive Supranuclear Palsy; Corticobasal Syndrome; Corticobasal Syndrome(CBS); Corticobasal Degeneration Syndrome; Corticobasal Degeneration; Corticobasal Degeneration (CBD); Corticobasal Syndrome (CBS); MSA; MSA - Multiple System Atrophy; MSA-C; Multiple System Atrophy; Multiple System Atrophy (MSA) With Orthostatic Hypotension; Multiple System Atrophy - Cerebellar Subtype (MSA-C); Multiple System Atrophy - Parkinsonian Subtype (MSA-P); Multiple System Atrophy, Cerebellar Type; Multiple System Atrophy, Parkinsonian Type; Progressive Supranuclear Palsy; Progressive Supranuclear Palsy(PSP); Progressive Supranuclear Palsy (PSP)
Keywords: genetic study; Progressive Supranuclear Palsy; Multiple System Atrophy; Corticobasal; CurePSP; PSP; MSA; CBD; Genes
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Shy-Drager Syndrome; Multiple System Atrophy; Multiple system atrophy (MSA) with orthostatic hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA from whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CurePSP Genetics Program: Adults with PSP, CBD or MSA
  Interventions: Other: Whole genome sequencing will be performed at the NIH

INTERVENTIONS:
Other: Whole genome sequencing will be performed at the NIH — All samples will undergo non-CLIA approved whole genome sequencing on a research basis in collaboration with Sonja Scholz, MD, PhD at the Neurodegenerative Diseases Research Unit of the National Institutes of Health (Bethesda, MD). This sequencing method allows for the identification of not only variants known to be associated with these disorders but also potentially novel variants.

SUMMARY:
This study is an observational, prospective genetic study. It aims to obtain DNA for research and testing from patients with PSP, CBS, MSA, and related neurological conditions and their families.

Up to 1,000 adults who have been clinically diagnosed with PSP, CBS, MSA, or related neurological conditions will be enrolled. The study intervention involves sequencing of participant blood samples using non-CLIA-approved whole genome sequencing at the National Institutes of Health. Pathogenic variants that are deemed possibly related to these conditions will be confirmed using CLIA-approved testing. The study involves minimal risk to participants.

DETAILED DESCRIPTION:
Genetic research is important for basic, translational, and clinical researchers, and are particularly important for rare disease investigations. Understanding a patient's genetic background may also facilitate participant recruitment for targeted genetic therapeutic trials and has the potential to empower participants with PSP, CBS, MSA, or related neurological diseases and clinicians to make more informed decisions about their clinical care plan. Furthermore, genetic research augments the clinical counseling process by offering participants and their families a clearer understanding of disease risk in relatives. Overall, this study may help to refine current diagnostic criteria for PSP, CBS, MSA, and related neurological conditions, inform genetic counseling, fuel future research studies, and provide insights into potential therapeutic paradigms.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged 35 or older) with a clinical diagnosis of PSP, CBS, MSA, or a related neurological disease as confirmed by their healthcare provider, or unaffected family members of participants who have reported a family history of relevant neurodegenerative conditions.
2. Meet Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Possible or Probable PSP (32), clinically established or clinically probable MSA (33), Armstrong criteria (2013) for possible or probable CBS (34). Diagnostic certainty will be determined by the treating/referring clinician.
3. Willingness to undergo genetic testing. Participants will have the option to receive relevant genetic test results.
4. Have the capacity to give full informed consent in writing or electronically, or provide consent through a legally authorized representative (LAR)/power of attorney (POA), and have read, understood, and completed the informed consent form.
5. Are able to perform or have a designee who can perform study activities (including completion of either online or orally administered surveys).

Exclusion Criteria:

1. Individuals who have received a blood transfusion within the past 3 months.
2. Individuals who have active hematologic malignancies such as lymphoma or leukemia.
3. Individuals who have had a bone marrow transplant within the past 5 years.
4. Individuals under the age of 35 or age of majority in applicable states at the time of consenting.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with PSP, CBD/CBS or MSA
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole genome sequencing | 5 years
  All samples will first undergo non-CLIA approved whole genome sequencing on a research basis in collaboration with Sonja Scholz, MD, PhD at the Neurodegenerative Diseases Research Unit of the National Institutes of Health (Bethesda, MD). This sequencing method allows for the identification of not only variants known to be associated with these disorders but also potentially novel variants.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All sequencing data will be deposited on a controlled-access repository such as the NIH Database of Genotypes and Phenotypes (dbGaP) and the Accelerating Medicines Partnership in Parkinson's Disease (AMP-PD) cloud-based data repository for data sharing by the genetic testing laboratory. Data access requests will be reviewed and approved by the corresponding repository's data access committee, such as the dbGaP Data Access Committee and the AMP-PD Access and Compliance Team, in accordance with their data use policies. No identifiable information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: June, 2025- December 2030
Access Criteria: Data access requests will be reviewed and approved by the corresponding repository's data access committee, such as the dbGAP Data Access Committee and the AMP-PD Access and Compliance Team, in accordance with their data use policies. No identifiable information will be shared.
URL: https://www.amp-pd.org/

REFERENCES:
- [Background] Jabbari E, Koga S, Valentino RR, Reynolds RH, Ferrari R, Tan MMX, Rowe JB, Dalgard CL, Scholz SW, Dickson DW, Warner TT, Revesz T, Hoglinger GU, Ross OA, Ryten M, Hardy J, Shoai M, Morris HR; PSP Genetics Group. Genetic determinants of survival in progressive supranuclear palsy: a genome-wide association study. Lancet Neurol. 2021 Feb;20(2):107-116. doi: 10.1016/S1474-4422(20)30394-X. Epub 2020 Dec 17. PMID 33341150
- [Background] Chen JA, Chen Z, Won H, Huang AY, Lowe JK, Wojta K, Yokoyama JS, Bensimon G, Leigh PN, Payan C, Shatunov A, Jones AR, Lewis CM, Deloukas P, Amouyel P, Tzourio C, Dartigues JF, Ludolph A, Boxer AL, Bronstein JM, Al-Chalabi A, Geschwind DH, Coppola G. Joint genome-wide association study of progressive supranuclear palsy identifies novel susceptibility loci and genetic correlation to neurodegenerative diseases. Mol Neurodegener. 2018 Aug 8;13(1):41. doi: 10.1186/s13024-018-0270-8. PMID 30089514
- [Background] Hoglinger GU, Melhem NM, Dickson DW, Sleiman PM, Wang LS, Klei L, Rademakers R, de Silva R, Litvan I, Riley DE, van Swieten JC, Heutink P, Wszolek ZK, Uitti RJ, Vandrovcova J, Hurtig HI, Gross RG, Maetzler W, Goldwurm S, Tolosa E, Borroni B, Pastor P; PSP Genetics Study Group; Cantwell LB, Han MR, Dillman A, van der Brug MP, Gibbs JR, Cookson MR, Hernandez DG, Singleton AB, Farrer MJ, Yu CE, Golbe LI, Revesz T, Hardy J, Lees AJ, Devlin B, Hakonarson H, Muller U, Schellenberg GD. Identification of common variants influencing risk of the tauopathy progressive supranuclear palsy. Nat Genet. 2011 Jun 19;43(7):699-705. doi: 10.1038/ng.859. PMID 21685912
- [Background] Rohrer JD, Paviour D, Vandrovcova J, Hodges J, de Silva R, Rossor MN. Novel L284R MAPT mutation in a family with an autosomal dominant progressive supranuclear palsy syndrome. Neurodegener Dis. 2011;8(3):149-52. doi: 10.1159/000319454. Epub 2010 Sep 14. PMID 20838030
- See also: Related Info — https://www.psp.org/genetic-program